CLINICAL TRIAL: NCT04708457
Title: A Pilot Feasibility RCT of Early ECMO to DE-sedate, Extubate, and Mobilise in Severe Acute Respiratory Infection
Brief Title: The REDEEM Pilot Study: A Feasibility RCT of Early ECMO in Severe Acute Respiratory Infection, Including COVID-19, WHO
Acronym: REDEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANZIC-RC/AB V3.1
Record Dates: First submitted 2020-12-04; First posted 2021-01-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Mechanical Ventilation Complication; Severe Acute Respiratory Infection; Covid19
Keywords: Intensive Care Unit; ECMO; Extracorporeal membrane oxygenation; Mechanical ventilation; Early ECMO
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early ECMO (Active Comparator): Early ECMO therapy for patients who have SARI and have been mechanically ventilated for 5-7 days.
  Interventions: Other: VV-ECMO
- Standard Care (No Intervention): Patients with SARI who are already mechanically ventilated will continue to receive the standard intensive care therapies, including ECMO if required.

INTERVENTIONS:
Other: VV-ECMO — Early use of VV-ECMO in SARI patients.
  Arms: Early ECMO

SUMMARY:
Patients who are critically ill in intensive care with moderate to severe acute respiratory infection often require mechanical ventilation. Prolonged ventilation increases the risk of lung damage and other side effects as a result of long term use of sedation medications. Extracorporeal membrane oxygenation therapy (ECMO), is a relatively new technology that uses a pump to remove blood from the body and return it back to the body after adding oxygen and removing carbon dioxide. ECMO can be used on patients who require mechanical ventilation and can function without the need for ongoing mechanical ventilation, thus reducing risk of side effects. Participants will be randomised into either the early ECMO therapy group or will continue standard treatment involving mechanical ventilation.

This pilot study aims to determine if a phase 3 Randomised Control Trial (RCT) is feasible for the use of early ECMO therapy to treat patients with Severe Acute Respiratory Infection (SARI). The success of the study will be determined by the successful recruitment of adult patients, that there is a difference between ECMO utilisation between groups and that there are no safety issues.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation is standard care for SARI and is associated with long term functional complications: Current guidelines recommend that mechanical ventilation, including protective lung strategies such as low tidal volumes, low peak pressures and titrated peak end expiratory pressure (PEEP), should form the mainstay of treatment for severe respiratory failure. While these strategies have been shown to reduce mortality, the application of invasive mechanical ventilation in the setting of SARIs may in fact propagate ongoing lung injury. Ventilator induced lung injury (VILI) results from the high pressures, over distension, and shear injury used by the ventilator to maintain gas exchange. Invasive ventilation can lead to secondary bacterial infection from poor clearance of sputum by sedated patients. And "air hunger" - the rapid and deep injurious breathing pattern by patients with severe lung injury - can lead to patient self-induced lung injury (P-SILI). Taken together, these factors can lead to a vicious cycle - the VILI Vortex - where lung damage leads to shrinkage of the functional lung unit, reduced compliance, higher transpulmonary pressures, worsening inflammation, further shrinkage, and ultimately even more severe lung damage and gas exchange failure.

Current strategies to facilitate mechanical ventilation include prolonged heavy sedation to assist patient-ventilator synchronization, and neuromuscular blockade (to prevent any spontaneous respiratory effort), often for weeks at a time. These interventions, plus the underlying lung damage, contribute to significant long term complications, including immobility and ICU myopathy, delirium, respiratory muscle weakness and tracheostomy, leading to significant delays in ICU and hospital discharge, rehabilitation, and return to home. Survivors of prolonged mechanical ventilation have been shown to have high rates of functional disability, immobility, psychological injury, and reduced health related quality of life - and these outcomes can persist for up to 5 years.

Thus, conventional treatment with mechanical ventilation, deep sedation, and/or neuromuscular paralysis is likely to adversely impact long term functional outcomes in patients with SARI. There is a clear unmet need for novel strategies that facilitate safe lung ventilation, while also limiting the intensity and duration of these interventions and complications.

ECMO is an external machine that oxygenates the blood in addition to a mechanical ventilator. Venous cannulae drain blood out of the body and return it back after an oxygenator adds oxygen and removes carbon dioxide. Venovenous (VV) ECMO supports patients with respiratory failure, by providing the body with sufficient oxygen and by removing all the carbon dioxide (CO2) in the blood (causing a respiratory alkalosis), which reduces the drive to breathe and permits "lung rest". Resting the lungs avoids VILI, reduces pulmonary and systemic inflammation, and reduces extra-pulmonary organ dysfunction. Traditionally, ECMO was employed very late in the course of the disease as a "rescue therapy", when patients already had severely damaged lungs, due to fears of complications such as bleeding that would worsen the patients multi organ failure. However advances in modern ECMO technology mean it is associated with a lower complication rate (<10% cannula site bleeding) and its use has doubled over the last five years. ECMO now offers the ideal platform to prevent ventilator-induced lung damage in patients that are less severely unwell, and earlier in the disease process, while also reducing the need for heavy sedation and/or neuromuscular blockade. It facilitates safe de-sedation without VILI as well as extubation, and physiotherapy-which is difficult to carry out adequately when a patient is sedated and ventilated. All these factors have been associated with improved long term health outcomes for patients.

This study aims to determine if a large RCT looking at use of early ECMO to treat patients with SARI is feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory confirmed severe acute respiratory infection (SARI) pneumonitis such as Coronavirus disease of 2019 (COVID-19) or influenza, AND
2. ≥5 days of mechanical ventilation, AND
3. Moderate to severe respiratory failure as shown by either the ratio of partial pressure of oxygen and the fracture of inspired oxygen (PaO2:FiO2 Rati)o <150 for >6 hours OR the potential of hydrogen (pH) <7.30 with carbon dioxide (CO2) >50mmHg for 6 hours, AND
4. Are unable to pass a spontaneous breathing trial.

Exclusion Criteria:

1. Age ≥70 year old
2. Extubation likely in next 24-48 hours
3. Duration of mechanical ventilation ≥7days
4. ≥2 non-pulmonary organ failures (as scored by the sequential oxygen failure assessment (SOFA) score)
5. Need for immediate VV ECMO (as per EOLIA (research study) criteria*)
6. Requirement for VA ECMO
7. Clinical frailty or ≥2 major comorbidities
8. The physician deems the study is not in the patient's interest

   * EOLIA criteria (P:F <50 for 3 hours, P:F<80 for 6 hours, pH<7.25 with carbon dioxide partial pressure (PCO2) >60 for >6 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who have SARI and have been mechanically ventilated for at least 5 days. | 12 months
  The number of participants who have SARI and have been mechanically ventilated for at least 5 days but no more than 7 days are eligible to participate in this study. The number of patients that meet this criteria will help assess the feasibility of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Burrell, MBBS, Principal Investigator — The Alfred
Locations (2):
- The Alfred Hospital, Melbourne, Victoria, Australia
- Charite Universitatmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No